CLINICAL TRIAL: NCT05554406
Title: A Randomized Phase II Study Comparing Cytarabine + Daunorubicin (7+3) vs (Daunorubicin and Cytarabine) Liposome, Cytarabine + Daunorubicin + Venetoclax, Azacitidine + Venetoclax, and (Daunorubicin and Cytarabine) Liposome + Venetoclax in Patients Aged 59 or Younger Who Are Considered High-Risk (Adverse) Acute Myeloid Leukemia As Determined by MYELOMATCH; A MYELOMATCH Clinical Trial
Brief Title: Testing the Effects of Novel Therapeutics for Newly Diagnosed, Untreated Patients With High-Risk Acute Myeloid Leukemia (A MyeloMATCH Treatment Trial)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-07535; NCI-2022-07535 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MM1YA-S01 (Other: SWOG); MM1YA-S01 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2022-09-22; First posted 2022-09-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia; Acute Myeloid Leukemia Arising From Previous Myelodysplastic/Myeloproliferative Neoplasm; Acute Myeloid Leukemia Post Cytotoxic Therapy; Acute Myeloid Leukemia, Myelodysplasia-Related
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myeloproliferative Disorders | interventions — Azacitidine; Specimen Handling; Cytarabine; Daunorubicin; CPX-351; Injections; Liposomes; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Arm I (cytarabine, daunorubicin) (Active Comparator): Patients receive cytarabine IV continuously on days 1-7 and daunorubicin IV on days 1-3 per standard approach of each cycle. Cycles repeat every 28 days for 1 cycle in the absence of disease progression or unacceptable toxicity. Patients may receive an additional cycle of cytarabine IV continuously on days 1-5 and daunorubicin IV on days 1-2. Patients undergo ECHO or MUGA scan during screening. Patients also undergo a bone marrow aspiration and collection of blood throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan
- Arm II (cytarabine, daunorubicin, venetoclax) (Experimental): Patients receive cytarabine IV continuously on days 2-8 and daunorubicin IV on days 2-4 with venetoclax PO on days 1-11 of each cycle. Cycles repeat every 28 days for 1 cycle in the absence of disease progression or unacceptable toxicity. Patients may receive an additional cycle of cytarabine IV continuously on days 2-6 and daunorubicin IV on days 2-3 with venetoclax PO on days 1-8. Patients undergo ECHO or MUGA scan during screening. Patients also undergo a bone marrow aspiration and collection of blood throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Drug: Venetoclax
- Arm III (azacitidine, venetoclax) (Experimental): Patients receive azacitidine SC or IV on days 1-7 and venetoclax PO on days 1-28 of each cycle. Cycles repeat every 28 days for 2 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO or MUGA scan during screening. Patients also undergo a bone marrow aspiration and collection of blood throughout the trial.
  Interventions: Drug: Azacitidine; Procedure: Biospecimen Collection; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Drug: Venetoclax
- Arm IV (daunorubicin and cytarabine liposome) (Experimental): Patients receive daunorubicin and cytarabine liposome IV over 90 minutes on days 1, 3, and 5 of each cycle. Cycles repeat every 28 days for 1 cycle in the absence of disease progression or unacceptable toxicity. Patients may receive an additional cycle of daunorubicin and cytarabine liposome IV over 90 minutes on days 1 and 3. Patients undergo ECHO or MUGA scan during screening. Patients also undergo a bone marrow aspiration and collection of blood throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Echocardiography Test; Drug: Liposome-encapsulated Daunorubicin-Cytarabine; Procedure: Multigated Acquisition Scan
- Arm V (daunorubicin and cytarabine liposome, venetoclax) (Experimental): Patients receive daunorubicin and cytarabine liposome IV over 90 minutes on days 1, 3, and 5 and venetoclax PO on days 1-14 of each cycle. Cycles repeat every 28 days for 1 cycle in the absence of disease progression or unacceptable toxicity. Patients may receive an additional cycle of daunorubicin and cytarabine liposome IV over 90 minutes on days 1 and 3 and venetoclax PO on days 1-7. Patients undergo ECHO or MUGA scan during screening. Patients also undergo a bone marrow aspiration and collection of blood throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Echocardiography Test; Drug: Liposome-encapsulated Daunorubicin-Cytarabine; Procedure: Multigated Acquisition Scan; Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine — Given SC or IV
  Other Names: 5 AZC; 5-AC; 5-Azacitidine; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
  Arms: Arm III (azacitidine, venetoclax)
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
  Arms: Arm I (cytarabine, daunorubicin); Arm II (cytarabine, daunorubicin, venetoclax); Arm IV (daunorubicin and cytarabine liposome); Arm V (daunorubicin and cytarabine liposome, venetoclax)
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
  Arms: Arm I (cytarabine, daunorubicin); Arm II (cytarabine, daunorubicin, venetoclax)
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
  Arms: Arm I (cytarabine, daunorubicin); Arm II (cytarabine, daunorubicin, venetoclax)
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Drug: Liposome-encapsulated Daunorubicin-Cytarabine — Given IV
  Other Names: CPX 351; CPX-351; CPX351; Cytarabine and Daunorubicin Liposomal; Cytarabine-Daunorubicin Liposome for Injection; Daunorubicin and Cytarabine (Liposomal); Liposomal AraC-Daunorubicin CPX-351; Liposomal Cytarabine-Daunorubicin; Liposome-encapsulated Combination of Daunorubicin and Cytarabine; Vyxeos
  Arms: Arm IV (daunorubicin and cytarabine liposome); Arm V (daunorubicin and cytarabine liposome, venetoclax)
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Venetoclax — Given PO
  Other Names: ABT 199; ABT-0199; ABT-199; ABT199; GDC 0199; GDC-0199; GDC0199; RG7601; Venclexta; Venclyxto
  Arms: Arm II (cytarabine, daunorubicin, venetoclax); Arm III (azacitidine, venetoclax); Arm V (daunorubicin and cytarabine liposome, venetoclax)

SUMMARY:
This phase II MyeloMATCH treatment trial tests whether the standard approach of cytarabine and daunorubicin in comparison to the following experimental regimens works to shrink cancer in patients with high risk acute myeloid leukemia (AML): 1) daunorubicin and cytarabine liposome alone; 2) cytarabine and daunorubicin with venetoclax; 3) azacitidine and venetoclax; 4) daunorubicin and cytarabine liposome and venetoclax. "High-risk" refers to traits that have been known to make the AML harder to treat. Cytarabine is in a class of medications called antimetabolites. It works by slowing or stopping the growth of cancer cells in the body. Daunorubicin is in a class of medications called anthracyclines. It also works by slowing or stopping the growth of cancer cells in the body. Azacitidine is in a class of medications called demethylation agents. It works by helping the bone marrow to produce normal blood cells and by killing abnormal cells. Venetoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. It may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. There is evidence that these newer experimental treatment regimens may work better in getting rid of more AML compared to the standard approach of cytarabine and daunorubicin.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare measurable residual disease (MRD) negative complete remission (CR) rates between each of the experimental regimens and cytarabine + daunorubicin (7+3).

SECONDARY OBJECTIVES:

I. To estimate the frequency and severity of toxicities with each of the regimens.

II. To estimate complete remission (CR) rates, complete remission with incomplete count recovery (CRi, with and without MRD) rates, event-free survival (EFS), time to relapse, relapse-free survival (RFS), and overall survival (OS) with each of the regimens.

III. To describe and compare MRD negative CR rates by genomic subgroups within and across randomized arms.

BANKING OBJECTIVE:

I. To bank specimens for future correlative studies.

OUTLINE: Patients are randomized to 1 of 5 arms.

ARM I: Patients receive cytarabine intravenously (IV) continuously on days 1-7 and daunorubicin IV on days 1-3 per standard approach of each cycle. Cycles repeat every 28 days for 1 cycle in the absence of disease progression or unacceptable toxicity. Patients may receive an additional cycle of cytarabine IV continuously on days 1-5 and daunorubicin IV on days 1-2. Patients undergo echocardiography (ECHO) or multigated acquisition (MUGA) scan during screening. Patients also undergo a bone marrow aspiration and collection of blood throughout the trial.

ARM II: Patients receive cytarabine IV continuously on days 2-8 and daunorubicin IV on days 2-4 with venetoclax orally (PO) on days 1-11 of each cycle. Cycles repeat every 28 days for 1 cycle in the absence of disease progression or unacceptable toxicity. Patients may receive an additional cycle of cytarabine IV continuously on days 2-6 and daunorubicin IV on days 2-3 with venetoclax PO on days 1-8. Patients undergo ECHO or MUGA scan during screening. Patients also undergo a bone marrow aspiration and collection of blood throughout the trial.

ARM III: Patients receive azacitidine subcutaneously (SC) or IV on days 1-7 and venetoclax PO on days 1-28 of each cycle. Cycles repeat every 28 days for 2 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO or MUGA scan during screening. Patients also undergo a bone marrow aspiration and collection of blood throughout the trial.

ARM IV: Patients receive daunorubicin and cytarabine liposome IV over 90 minutes on days 1, 3, and 5 of each cycle. Cycles repeat every 28 days for 1 cycle in the absence of disease progression or unacceptable toxicity. Patients may receive an additional cycle of daunorubicin and cytarabine liposome IV over 90 minutes on days 1 and 3. Patients undergo ECHO or MUGA scan during screening. Patients also undergo a bone marrow aspiration and collection of blood throughout the trial.

ARM V: Patients receive daunorubicin and cytarabine liposome IV over 90 minutes on days 1, 3, and 5 and venetoclax PO on days 1-14 of each cycle. Cycles repeat every 28 days for 1 cycle in the absence of disease progression or unacceptable toxicity. Patients may receive an additional cycle of daunorubicin and cytarabine liposome IV over 90 minutes on days 1 and 3 and venetoclax PO on days 1-7. Patients undergo ECHO or MUGA scan during screening. Patients also undergo a bone marrow aspiration and collection of blood throughout the trial.

After completion of study treatment, patients follow up every month for the first year, every 2 months for the second year, every 3 months for the third year and every 6 months to year 5.

ELIGIBILITY:
Inclusion Criteria:

* STEP 1 REGISTRATION:
* Participants must have been registered to Master Screening and Re-Assessment Protocol, MYELOMATCH, prior to consenting to this study. Participants must have been assigned to this clinical trial, via MATCHBox, prior to registration to this study.

  * Note: Pre-enrollment/diagnosis labs must have already been performed under MYELOMATCH
* Participants must have newly diagnosed, untreated acute myeloid leukemia (AML) per World Health Organization (WHO) criteria
* Participants must have high-risk (adverse) AML per European LeukemiaNet (ELN) 2017 criteria
* Participants with therapy-related AML (t-AML), or with AML evolving from an antecedent hematologic disorder (such as myeloproliferative neoplasm), or AML with myelodysplasia-related changes (AML-MRC) are eligible
* Acute promyelocytic leukemia is excluded
* Participants with favorable or intermediate risk disease are excluded
* Participants with FLT3 mutations (ITD or TKD) are excluded
* Participants with t(9;22) translocation are excluded
* A single dose of intrathecal chemotherapy is allowed prior to study entry
* Prior anthracycline therapy is allowed but must not exceed a cumulative lifetime dose of 200 mg/m^2 daunorubicin or equivalent. Prior hypomethylating agent (HMA) exposure is allowed, as long as not for AML diagnosis
* Participants must not have received or be currently receiving any prior therapy for acute myeloid leukemia. Hydroxyurea to control the white blood cells (WBC) is allowed prior to registration and initiation of protocol-defined therapy. All trans retinoic acid (ATRA) given until a diagnosis of acute promyelocytic leukemia is ruled out is also allowed.
* Participants must not be receiving or planning to receive any other investigational agents before completing protocol therapy
* Participants must be between 18 and 59 years of age
* Participants must have Zubrod performance status =< 3 as determined by a history and physical (H&P) completed within 14 days prior to registration
* Participants must have a complete medical history and physical exam within 7 days prior to registration
* Participants must be able to swallow and retain oral medications and have no known gastrointestinal disorders likely to interfere with absorption of oral medications
* Participants with known human immunodeficiency virus (HIV)-infection must be on effective anti-retroviral therapy at time of registration and have undetectable HIV viral load within 6 months prior to registration
* Participants with evidence of chronic hepatitis B virus (HBV) infection must have undetectable HBV viral load within 28 days prior to registration and be on suppressive therapy, if indicated
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. Participants with active HCV infection who are currently on treatment must have an undetectable HCV viral load within 28 days prior to registration
* The following tests must be performed within 14 days prior to registration to establish baseline values:

  * Complete blood count (CBC)/differential/platelets
  * Total bilirubin
  * Lactate dehydrogenase (LDH)
  * Albumin
  * Glucose
  * Fibrinogen
* Participants must have adequate kidney function as evidenced by creatinine clearance >= 30mL/min (by Cockcroft Gault) within 28 days prior to registration
* Participants must have adequate liver function as evidenced by aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3.0 x upper limit of normal (ULN) within 28 days prior to registration
* Total bilirubin =< 2.0 x ULN (or 5.0 x ULN if the participant has a history of Gilbert's disease) within 28 days prior to registration
* Participants must have adequate cardiac function as determined by echocardiography or MUGA scan with an ejection fraction >= 50% within 28 days prior to registration
* Participants with a prior or concurrent malignancy whose natural history (in the opinion of the treating physician) does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial. No concurrent therapies for such malignancy are allowed with the exception of hormonal therapy
* Participants with known history of Wilson's disease or other known copper-metabolism disorder are excluded
* Participants must not be pregnant or nursing. Women/men of reproductive potential must have agreed to use 2 contraception methods. A woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months. In addition to routine contraceptive methods (e.g., hormonal contraceptives [examples include birth control pills, vaginal rings, or patches] associated with inhibition of ovulation for at least 1 month prior to taking study drug), "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation. However, if at any point a previously celibate participant chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures. A barrier method should be used during this study along with hormonal contraceptives from initial study drug administration to 30 days after the last dose of study drug as drug-drug interaction with venetoclax is unknown
* Participants must have agreed to have specimens submitted for translational medicine (MRD) under the myeloMATCH MSRP and specimens must be submitted
* Participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 335 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Minimal residual disease (MRD) response (Arm 1, 2, 4 and 5) | After induction (28 days) or re-induction (56 days)
  Will be analyzed using intent-to-treat (ITT) principles.
MRD response (Arm 3) | After two cycles of therapy (56 days)
  Will be analyzed using ITT principles.

SECONDARY OUTCOMES:
Early mortality | On or before day 28
  Will be assessed by death due to any cause between experimental arms and the 7+3 arm will be reported for each arm every data and safety monitoring committee (DSMC) cycle. Fisher's exact will be used to compare observed rates. A one-sided p-value < 0.05 indicating increased early mortality rates in an experimental arm will be a threshold for termination of accrual to an arm due to increased early mortality.
Time to count recovery | After cycle 1 and cycle 2
  Will be reported every DSMC cycle for the 7+3+venetoclax, (daunorubicin and cytarabine) liposome+venetoclax, and 7+3 arms. Median time to count recovery more than 7 days longer on either of the 7+3+venetoclax and (daunorubicin and cytarabine liposome+venetoclax arms compared to the 7+3 arm will be used a threshold to terminate accrual to an arm due to increased toxicity.
Event-free survival | From randomization to the first of: primary refractory disease; progressive disease; off protocol therapy without complete remission (CR) or CR with incomplete count recovery (CRi); relapse from CR or CRi, or death from any cause, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method.
Relapse-free survival | From the date of achievement of a remission until the date of relapse or death from any cause, assessed up to 5 years
  Defined for only patients achieving CR, or CRi. Will be estimated using the Kaplan-Meier method.
Overall survival | From day of randomization on study until death from any cause, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method.
Time to relapse | Up to 5 years
  Will be estimated with cumulative incidence curves with death without relapse analyzed a competing event. Response per 2017 European LeukemiaNet guidelines will be tabulated and exact 95% confidence intervals will be calculated.
MRD negative complete remission (MRDneg CR) | Up to 5 years
  MRDneg CR rates will be tabulated by genomic subgroups within randomized arms and pooling arms. Rates across arms will be compared using Fisher's exact test. All p-values reported will be nominal.
Incidence of adverse events | Up to 5 years
  Will be analyzed using National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Shami, Principal Investigator — SWOG Cancer Research Network
Locations (203):
- United States (196):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Mills Health Center, San Mateo, California
  - Yale University, New Haven, Connecticut
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - UChicago Medicine Northwest Indiana, Crown Point, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Our Lady of The Lake, Baton Rouge, Louisiana
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Lahey Medical Center-Peabody, Peabody, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Mount Sinai Hospital, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - ThedaCare Regional Medical Center - Appleton, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- Canada (5):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - QEII Health Sciences Centre/Nova Scotia Health Authority, Halifax, Nova Scotia
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
- Puerto Rico (2):
  - Centro Comprensivo de Cancer de UPR, San Juan
  - San Juan City Hospital, San Juan

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm